CLINICAL TRIAL: NCT03756948
Title: Association Between Viscoelastic Tests-Guided Therapy With Synthetic Factor Concentrates And Allogenic Blood Transfusion In Liver Transplantation: A Before-After Study
Brief Title: Viscoelastic Tests-Guided Therapy In Liver Transplantation
Acronym: VETLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VETLT
Record Dates: First submitted 2018-11-16; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Liver Transplant; Complications; Bleeding; Hemostatic Disorder
Keywords: Liver Transplantation; Blood Coagulation Disorders; Blood Transfusion; Hemostasis; Thromboelastometry
MeSH Terms: conditions — Hemorrhage; Hemostatic Disorders; Blood Coagulation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Before) (Active Comparator): No Thromboelastometry No Synthetic Factor Concentrates Usual Care
  Interventions: Other: Usual Care
- Thromboelastometry-Guided Therapy (After) (Experimental): Thromboelastometry-Guided Therapy with Synthetic Factor Concentrates
  Interventions: Other: Thromboelastometry-Guided Therapy with Synthetic Factor Concentrates

INTERVENTIONS:
Other: Usual Care — Treatment of Coagulation Disorders Using Standard Coagulation Tests and Blood Components
  Arms: Usual Care (Before)
Other: Thromboelastometry-Guided Therapy with Synthetic Factor Concentrates — Thromboelastometry-Guided Treatment of Coagulation Disorders Using Synthetic Factor Concentrates
  Arms: Thromboelastometry-Guided Therapy (After)

SUMMARY:
BACKGROUND: Perioperative bleeding and transfusion are important causes of morbidity and mortality in patients undergoing liver transplantation. The aim of this study is to assess whether viscoelastic tests-guided therapy with the use of synthetic factor concentrates impact transfusion rates of hemocomponents in adult patients undergoing liver transplantation.

METHODS: This is an interventional before-after comparative study. Patients undergoing liver transplantation before the implementation of a protocol using thromboelastometry and synthetic factor concentrates were compared to patients after the implementation. Primary outcome was transfusion of any hemocomponents. Secondary outcomes included: transfusion of red blood cells (RBC), fresh frozen plasma (FFP), cryoprecipitate or platelets, clinical complications, length of stay and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Deceased Donor Liver Transplantation
* Chronic Liver Disease

Exclusion Criteria:

* Acute Liver Failure
* Combined Transplantation
* Re-Transplantation is Less Than 30 Days After the First Transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Need of Any Blood Products Transfusion | 48 Hours
  Collapsed composite of need of any transfusion of blood product during surgery and in the first 48 hours in the postoperative, including the need of RBC, FFP, cryoprecipitate and/or platelets.

SECONDARY OUTCOMES:
Use of Synthetic Factor Concentrates or Antifibrinolytic | 48 Hours
  Any use of synthetic factor concentrates or antifibrinolytic
Clinical Complications Related to the Procedure | Third days or until hospital discharge, whichever occurs first
  Defined as: 1) Upper digestive hemorrhage; 2) Arterial thrombosis; 3) Infection; and/or 4) Any thromboembolic event
Duration of Mechanical Ventilation | Third days or until hospital discharge, whichever occurs first
  Duration of mechanical ventilation in the post-operative period
ICU Length of Stay | Third days or until ICU discharge, whichever occurs first
  Duration of stay in the intensive care unit
Hospital Length of Stay | Third days or until hospital discharge, whichever occurs first
  Duration of stay in the hospital
In-Hospital Mortality | Third days or until hospital discharge, whichever occurs first
  Any death during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ary Serpa Neto, MD, MSc, PhD, Principal Investigator — Physician and Researcher; Raffael PC Zamper, MD, Study Director — Raffael

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rana A, Petrowsky H, Hong JC, Agopian VG, Kaldas FM, Farmer D, Yersiz H, Hiatt JR, Busuttil RW. Blood transfusion requirement during liver transplantation is an important risk factor for mortality. J Am Coll Surg. 2013 May;216(5):902-7. doi: 10.1016/j.jamcollsurg.2012.12.047. Epub 2013 Mar 9. PMID 23478547
- [Background] Hartmann M, Szalai C, Saner FH. Hemostasis in liver transplantation: Pathophysiology, monitoring, and treatment. World J Gastroenterol. 2016 Jan 28;22(4):1541-50. doi: 10.3748/wjg.v22.i4.1541. PMID 26819521
- [Background] Luddington RJ. Thrombelastography/thromboelastometry. Clin Lab Haematol. 2005 Apr;27(2):81-90. doi: 10.1111/j.1365-2257.2005.00681.x. PMID 15784122
- [Background] Weber CF, Gorlinger K, Meininger D, Herrmann E, Bingold T, Moritz A, Cohn LH, Zacharowski K. Point-of-care testing: a prospective, randomized clinical trial of efficacy in coagulopathic cardiac surgery patients. Anesthesiology. 2012 Sep;117(3):531-47. doi: 10.1097/ALN.0b013e318264c644. PMID 22914710
- [Background] Wang SC, Shieh JF, Chang KY, Chu YC, Liu CS, Loong CC, Chan KH, Mandell S, Tsou MY. Thromboelastography-guided transfusion decreases intraoperative blood transfusion during orthotopic liver transplantation: randomized clinical trial. Transplant Proc. 2010 Sep;42(7):2590-3. doi: 10.1016/j.transproceed.2010.05.144. PMID 20832550
- [Derived] Zamper RPC, Amorim TC, Queiroz VNF, Lira JDO, Costa LGV, Takaoka F, Juffermans NP, Neto AS. Association between viscoelastic tests-guided therapy with synthetic factor concentrates and allogenic blood transfusion in liver transplantation: a before-after study. BMC Anesthesiol. 2018 Dec 22;18(1):198. doi: 10.1186/s12871-018-0664-8. PMID 30579327